CLINICAL TRIAL: NCT06063447
Title: Relationship Between the Type and Severity of Scoliosis and Pelvic Floor Dysfunctions in Individiuals With Adolescent Idiopathic Scoliosis
Brief Title: Does Adolescent Idıopathic Scoliosis Cause Pelvic Floor Dysfunction?
Status: Completed | Type: Observational
Sponsor: Cyprus International University (Other)
Collaborators: Near East University, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: 020-6029
Record Dates: First submitted 2023-09-21; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Scoliosis Idiopathic; Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Floor Disorders | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Examination — Posture Evaluation, Scoliosis Examination, Pelvic Floor Assesments

SUMMARY:
The aim of this study was to investigate relationship between the type and severity of scoliosis and pelvic floor dysfunctions in individuals with adolescent idiopathic scoliosis.

DETAILED DESCRIPTION:
While a healthy spine has a flat appearance in the axial line in the frontal plane, individuals with scoliosis have lateral flexion to one side and rotation deformity in the horizantal plane. In other words, it is a 3-dimensional problem that causes severe postural disorder in advanced stages, accompanied by lateral flexion of the spine of 10 degrees or more in the frontal plane, axial rotation in the transverse plane and kyphosis-lordosis deformity in the sagittal plane. Especially the "core" region, which is formed by 4 main muscle groups, stabilizes the pelvic organs by balancing intra-abdominal pressure increases and provides spinal stabilization. Studies showing that pelvic floor functions may be affected in normal spinal physiologic curvature changes are available in the literature. However, the relationship between the angle and severity of scoliosis and pelvic floor dysfunctions due to idiopathic scoliosis has not been clearly clarified.

In this context, the study aims to evaluate and compare scoliosis-related parameters (type of scoliosis, cobb angle, axial rotation angle), pelvic floor dynamics and dysfunctions in individuals with idiopathic scoliosis and healthy individuals with the same age group and characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Those with adolescent idiopathic scoliosis diagnosed above 10' degree,
* Under 19 years of age diagnosed with AIS,
* Individuals whose consent was obtained from their families to participate in the study

Exclusion Criteria:

* Those with congenital scoliosis,
* Those with a history of neuromuscular disease,
* Diagnosed with any systemic disease other than AIS,
* Those with a history of malignancy and/or ongoing treatment,
* Those with a history of urogenital diseases and surgical history,
* Individuals with previous spinal surgery

Ages: 11 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Individuals aged between 11-18 years and followed up in physiotherapy centers that met the inclusion criteria were selected.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Scoliosis | 10 minutes
  With X-Ray
Posture Analysis | 5 minutes
  With Posture Screen Mobile Application
Pelvic Floor Muscle Activity | 15 Minutes
  With Real Time Transabdominal Ultrasound
Pelvic Floor Dysfunction | 5 minutes
  With Pelvic Floor Distress Inventory
Dysfunctional Voiding | 10 minutes
  With Dysfunctional Voiding Scoring System

CONTACTS AND LOCATIONS:
Overall Officials: Salih Angın, Prof., Study Chair — Cyprus International University
Locations (1):
- Batuhan Ibrahim, Mersin, Lefkosa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perkins, J., Boyer, A., Mcleish, A., & Grossnickle, K. (2012). Idiopathic scoliosis and pelvic floor dysfunction. International Journal of Therapy and Rehabilitation, 19(2), 106-110.
- [Background] Meyer I, McArthur TA, Tang Y, McKinney JL, Morgan SL, Richter HE. Pelvic Floor Symptoms and Spinal Curvature in Women. Female Pelvic Med Reconstr Surg. 2016 Jul-Aug;22(4):219-23. doi: 10.1097/SPV.0000000000000271. PMID 27054800
- [Background] Naziri Q, Detolla J, Hayes W, Burekhovich S, Merola A, Akamnanu C, Paulino CB. A Systematic Review of All Smart Phone Applications Specifically Aimed for Use as a Scoliosis Screening Tool. J Long Term Eff Med Implants. 2018;28(1):25-30. doi: 10.1615/JLongTermEffMedImplants.2017020737. PMID 29772989
- [Background] Negrini S, Donzelli S, Aulisa AG, Czaprowski D, Schreiber S, de Mauroy JC, Diers H, Grivas TB, Knott P, Kotwicki T, Lebel A, Marti C, Maruyama T, O'Brien J, Price N, Parent E, Rigo M, Romano M, Stikeleather L, Wynne J, Zaina F. 2016 SOSORT guidelines: orthopaedic and rehabilitation treatment of idiopathic scoliosis during growth. Scoliosis Spinal Disord. 2018 Jan 10;13:3. doi: 10.1186/s13013-017-0145-8. eCollection 2018. PMID 29435499
- [Background] Ahmed SA., Othman NA., Sabet NA., & Salwa F. (2021). Validity and Reliability of Posture Screen Mobile Application in Adolescent Idiopathic Scoliosis. The Medical Journal of Cairo University, 89(June), 737-743.